CLINICAL TRIAL: NCT06500234
Title: Phase III Study on the Relation of Nutrition and Immunotherapy of Cancer Patients
Brief Title: Nutrition Impact on Immunotherapy of Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qingdao Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY202400918
Record Dates: First submitted 2024-07-04; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Nutrition Disorders; Immunotherapy; Cancer; Survival, Prosthesis
MeSH Terms: conditions — Nutrition Disorders; Neoplasms; Prosthesis Failure | interventions — Megestrol Acetate; Olanzapine

STUDY DESIGN:
Intervention Model Description: Malnourished patients with megestrol acetate 160mg oral, olanzapine 2.5mg oral, everyday during the immunotherapy course or intolerable.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- megestrol acetate-olanzapine (Experimental): Megestrol acetate 160 mg, oral, everyday Olanzapine 2.5 mg, oral everyday
  Interventions: Drug: Megestrol Acetate and olanzapine
- control (Placebo Comparator): Starch powder 50 mg, oral, everyday,
  Interventions: Drug: Starch powder 50 mg

INTERVENTIONS:
Drug: Megestrol Acetate and olanzapine — megestrol acetate, 160 mg, oral everyday; olanzapine 2.5 mg, oral everyday
  Arms: megestrol acetate-olanzapine
Drug: Starch powder 50 mg — Starch powder 50 mg, oral, everyday
  Arms: control

SUMMARY:
This study investigates nutritional status and outcomes of immuntherapy in cancer patients.

DETAILED DESCRIPTION:
Studies have shown that more than half of the patients with cancer are also malnourished at diagnosis. This increases patients' risk of complications associated with the treatment as well as the abandonment of care, as well as decrease the level of survival rates.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer, malnutrition Age >18 years Performance status ECOG of 0 or 2. Life expectancy ≥ 6 months. At least one lesion measurable as defined by standard imaging criteria for the patient's tumor type (RECIST v1.1) Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment Postmenopausal or evidence of non-childbearing status for women of childbearing potential Patient is willing and able to comply with the protocol for the duration of the study.

For all oral medications patients must be able to comfortably swallow capsules;

Exclusion Criteria:

* Patients unable to swallow orally administered medication and patients with Impairment of gastrointestinal (GI) function or GI disease that may significantly alter drug absorption of oral drugs History of allogenic organ, bone marrow or double umbilical cord blood transplantation.

Active or prior documented autoimmune or inflammatory disorders Uncontrolled intercurrent illness or patient considered a poor medical risk due to a serious, uncontrolled medical disorder, including but not limited to, ongoing or active infection, symptomatic congestive heart failure Currently taking medications with known risk of prolonging the QT interval or inducing Torsades de Pointes.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 12 months
  overall response rate

SECONDARY OUTCOMES:
PFS | 12 months
  profression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: chunling zhang, MD, Study Chair — Qingdao Central Hospital
Locations (1):
- Qingdao Central Hospital, Qingdao, Shandong, China